CLINICAL TRIAL: NCT03855020
Title: Serial Epstein-Barr Virus DNA Surveillance During Treatment in Non-metastatic Nasopharyngeal Carcinoma Patients
Brief Title: Serial Epstein-Barr Virus DNA Surveillance in Nasopharyngeal Carcinoma Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ying Sun, Vice-president, Sun Yat-sen University
Other Study IDs: 2019-FXY-015-radiation
Record Dates: First submitted 2019-02-21; First posted 2019-02-26 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: plasma EBV DNA; nasopharyngeal carcinoma; longitudinal surveillance
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- observational cohort: Patients enrolled in this observational cohort would have regular blood taking for EBV DNA examination at baseline, after every cycle of chemotherapy, every week during radiotherapy, and 1-3 months after chemo-radiotherapy until EBV DNA becomes undetectable for at least two times.
  Interventions: Diagnostic Test: Plasma EBV DNA

INTERVENTIONS:
Diagnostic Test: Plasma EBV DNA — Parameters analyzed will include (1) the changing pattern of plasma EBV DNA concentrations during chemotherapy and radiotherapy (2) half-life values (t1/2) of plasma EBV DNA clearance rate

SUMMARY:
Endemic nasopharyngeal carcinoma (NPC) is invariably associated with Epstein-barr virus (EBV) infection. Plasma EBV DAN detected by polymerase chain reaction (PCR)-based assays can provide important informations of disease screening, disease relapse, and risks classification. In this study, the investigators will explore the impact of serial plasma EBV DNA during chemotherapy and radiotherapy on initial tumor response and long-term survival in patients with non-metastatic nasopharyngeal carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly histologically confirmed non-keratinizing carcinoma (according to WHO histological type)
2. No evidence of distant metastasis (M0)
3. Receive standard radical treatment
4. Not exhibiting overt psychopathology, and willing to participate and written informed consent was obtained

Exclusion Criteria:

1. WHO type keratinizing squamous cell carcinoma or basaloid squamous cell carcinoma.
2. Treatment with palliative intent
3. Previous chemotherapy or radiotherapy (except non-melanomatous skin cancers outside the intended RT treatment volume)
4. Severe intercurrent disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically confirmed, non-metastatic, previously untreated nasopharyngeal carcinoma (NPC) will be invited to join this study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-05-09 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 3 years
  Progression-free survival is calculated from the date of diagnosis of NPC to the date of progression of NPC or the date of death from any cause, whichever comes earlier.

SECONDARY OUTCOMES:
overall survival | 3 years
  Overall survival is calculated from the date of diagnosis of NPC to the date of death from any cause
Distant metastasis-free survival | 3 years
  Distant metastasis-free survival is calculated from the date of diagnosis of NPC to the date of distant metastasis or date of death from any cause, whichever comes earlier.
locoregional failure-free survival | 3 years
  Local or regional failure-free survival is calculated from the date of diagnosis of NPC to the date of regional nodal failure or date of death from any cause, whichever comes earlier.
EBV DNA clearance rate | during the first month
  The half-life value (t1/2) of plasma EBV DNA clearance was calculated using the equation of [t1/2 = 0.693/k].

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
not to share individual participant data (IPD) available to other researchers unless reasonably required, and only the PI has the whole access to the complete data